CLINICAL TRIAL: NCT02221388
Title: Relative Bioavailability of Different Salt Forms and Formulations of Single Doses Either 50 or 200 mg BI 671800 in the Fasted or Fed State. An Open-label, Randomised, Phase I Study With a 3-period Crossover Followed by Two Treatment Periods in Fixed Sequence in Healthy Male and Female Volunteers
Brief Title: Relative Bioavailability of Different Formulations of BI 671800 in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1268.56
Record Dates: First submitted 2014-08-19; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

ARMS (6):
- BI 671800 ED capsules (Active Comparator)
  Interventions: Drug: BI 671800 ED, 100 mg capsules
- BI 671800 HEA tablet in fasted state (Experimental)
  Interventions: Drug: BI 671800 HEA, 200 mg tablets
- BI 671800 HEA EC tablet in fasted state (Experimental)
  Interventions: Drug: BI 671800 HEA EC, 200 mg tablets
- BI 671800 HEA tablet in fed state (Experimental)
  Interventions: Drug: BI 671800 HEA, 200 mg tablets; Other: Standard meal
- BI 671800 HEA EC tablet in fed state (Experimental)
  Interventions: Drug: BI 671800 HEA EC, 200 mg tablets; Other: Standard meal
- BI 671800 HEA, 50 mg tablet in fasted state (Experimental)
  Interventions: Drug: BI 671800 HEA, 50 mg tablets

INTERVENTIONS:
Drug: BI 671800 HEA, 200 mg tablets
  Arms: BI 671800 HEA tablet in fasted state; BI 671800 HEA tablet in fed state
Drug: BI 671800 HEA EC, 200 mg tablets
  Arms: BI 671800 HEA EC tablet in fasted state; BI 671800 HEA EC tablet in fed state
Drug: BI 671800 HEA, 50 mg tablets
  Arms: BI 671800 HEA, 50 mg tablet in fasted state
Drug: BI 671800 ED, 100 mg capsules
  Arms: BI 671800 ED capsules
Other: Standard meal
  Arms: BI 671800 HEA EC tablet in fed state; BI 671800 HEA tablet in fed state

SUMMARY:
To compare the oral bioavailability and rate of absorption of two different formulations of BI 671800 HEA (choline salt) tablets 200 mg, one with enteric coating (EC) and one without EC, versus 2 x 100 mg BI 671800 ED (ethylenediamine salt) capsules. Both BI 671800 HEA formulations were further investigated concerning food effect and one of the two BI 671800 HEA formulations identified by interim pharmacokinetic analysis was further investigated concerning dose proportionality with 50 mg.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females according to the following criteria: Based upon a complete medical history, including physical examination, vital signs (BP, PR), 12-lead ECG, clinical laboratory tests
* Age 21 to 50 years (incl.)
* BMI 18.5 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with GCP and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy or hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs within one month or less than 10 half-lives of the respective drug prior to first study drug administration
* Participation in another trial with an investigational drug within 2 months prior to administration or during the trial
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes daily)
* Alcohol abuse (average consumption of more than 20 g/day in females and 30 g/day in males)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to day 1 of visit 2)
* Any laboratory value outside the reference range that is of clinical relevance, especially repeated alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyltransferase (GGT), alkaline phosphatase (ALP) or total bilirubin above upper limit of normal (ULN) at screening and not resolved before dosing.
* Inability to comply with dietary regimen of trial site
* Unwilling to avoid excessive sunlight exposure
* Use of drugs which might reasonably influence the results of the trial or that prolong the QT/QTc interval within 10 days prior to administration or during the trial, and CYP2C8 substrates such as amiodarone, amodiaquine, paclitaxel, rosiglitazone, pioglitazone and repaglinide or CYP2C9 such as warfarin, tolbutamide, phenytoin, losartan, acenocoumarol within 1 month or six half lives (whichever is greater).
* A marked baseline prolongation of the QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalaemia, family history of Long QT Syndrome)

For female subjects of childbearing potential only:

* Positive pregnancy test, pregnancy or planning to become pregnant during the study or within 2 months after study completion
* No adequate contraception during the study including three months before first dosing until 2 month after study completion, e.g. not any of the following: implants, injectables, combined hormonal contraceptives, intrauterine device, or surgical sterilisation (including hysterectomy). In addition to this, also a barrier method (e.g. condom) will be required, if the female is not surgically sterilised.
* Lactation

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum measured concentration of BI 671800 in plasma) | Up to 24 hours after last drug administration
AUC0-∞ (area under the concentration time curve of BI 671800 in plasma over the time interval from 0 extrapolated to infinity) | Up to 24 hours after last drug administration

SECONDARY OUTCOMES:
tmax (time from dosing to the maximum concentration of BI 671800 in plasma) | Up to 24 hours after last drug administration
AUC0-tz (area under the concentration-time curve of BI 671800 in plasma over the time interval from 0 to the time of the last quantifiable data point) | Up to 24 hours after drug administration
λz (terminal rate constant in plasma) | Up to 24 hours after drug adminnistration
t½ (terminal half-life of BI 671800 in plasma) | Up to 24 hours after drug administration
MRTpo (mean residence time of BI 671800 in the body after po administration) | Up to 24 hours after drug administration
CL/F (apparent clearance of BI 671800 in the plasma after extravascular administration) | Up to 24 hours after drug administration
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | Up to 24 hours after drug administration
Number of patients with clinical significant findings in physical examinations | Up to 10 days after last drug admininstration
Number of patients with clinical significant findings in vital signs | Up to 10 days after last drug administration
Number of patients with clinical significant findings in ECG | Up to 10 days after last drug administration
Number of patients with clinical significant findings in laboratory tests | Up to 10 days after last drug administration
Number of patients with adverse events | Up to 10 days after last drug administration
Investigator assessed tolerability on a 4 point scale | Up to 10 days after last drug administration